CLINICAL TRIAL: NCT04487457
Title: Étude Prospective d'évaluation de la cinétique Sanguine de Cellules Immunitaires et de Cytokines Immunosuppressives après Exposition à un Inhibiteur Des Checkpoints de l'immunité (ICI) : étude de l'Impact de la chimiothérapie
Brief Title: Prospective Study to Evaluate the Blood Kinetics of Immune Cells and Immunosuppressive Cytokines After Exposure to an Immunity Checkpoint Inhibitor (ICI): Study of the Impact of Chemotherapy
Acronym: CINECI
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI20 / CINECI; 2020-A01478-31 (Other: IdRCB)
Record Dates: First submitted 2020-07-16; First posted 2020-07-27 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer; Bladder Cancer; ENT Cancer
Keywords: Immunity checkpoint inhibitor; Rescue chemotherapy; Non Small Cell Lung Cancer; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer: Patients receiving chemotherapy alone after immunotherapy for NSCLC or bladder cancer or ENT cancer
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples

SUMMARY:
Non-small cell lung cancer (NSCLC) is the most common histological form, accounting for 85% of all bronchopulmonary cancers (PBC). The advent of Immunity Checkpoint Inhibitors (ICIs) targeting Programmed cell Death-1 (PD-1) is changing current treatment algorithms.

Preliminary results from work carried out in the Medical Oncology Department of the University Hospital of Tours suggest that immunotherapy targeting ICI, when administered beforehand, increases the effect of catch-up chemotherapy. In NSCLC, the progression-free survival (PFS) of 3rd line chemotherapy after anti-PD-1 immunotherapy was better than the PFS of 3rd line chemotherapy performed at the end of conventional chemotherapy. Moreover, the combination of chemotherapy and immunotherapy gives paradoxically better results than immunotherapy alone.

Immunotherapy restores the anti-tumor T immunity inhibited by the cancer cell. While the mode of action of ICIs is well known, the mechanisms of resistance to them are poorly understood. Several pathways are evoked, in particular the modulation of cellular interactions within the tumour microenvironment (TME), the molecular expression profile of cancer cells, or the immunological status of the patient.

Regulatory T lymphocytes (Treg) participate in the maintenance of immune system homeostasis by ensuring tolerance to self antigens. Within TME, Treg inhibit anti-tumor T cell activity and potentiate tumor proliferation. The latter, by specifically recognizing tumor antigens, block the activity of effector T lymphocytes directed against tumor cells. Thus, an increase in circulating Treg concentrations and in TME is a poor prognostic factor, especially in NSCLC.

Gemcitabine chemotherapy is commonly used in the management of NSCLC. Recent data show that gemcitabine decreases Treg activity and regulates levels of anti-inflammatory TME cytokines such as IL10, TGF-β and interferon-Ɣ.

The hypothesis of this study is that the decrease in Treg blood concentration by catch-up chemotherapy restores sensitivity to immunotherapy.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the most common histological form, accounting for 85% of all bronchopulmonary cancers (PBC). The advent of Immunity Checkpoint Inhibitors (ICIs) targeting Programmed cell Death-1 (PD-1) is changing current treatment algorithms.

Preliminary results from work carried out in the Medical Oncology Department of the University Hospital of Tours suggest that immunotherapy targeting ICI, when administered beforehand, increases the effect of catch-up chemotherapy. In NSCLC, the the progression-free survival (PFS) of 3rd line chemotherapy after anti-PD-1 immunotherapy was better than the PFS of 3rd line chemotherapy performed at the end of conventional chemotherapy. Moreover, the combination of chemotherapy and immunotherapy gives paradoxically better results than immunotherapy alone.

Immunotherapy restores the anti-tumor T immunity inhibited by the cancer cell. While the mode of action of ICIs is well known, the mechanisms of resistance to them are poorly understood. Several pathways are evoked, in particular the modulation of cellular interactions within the tumour microenvironment (TME), the molecular expression profile of cancer cells, or the immunological status of the patient.

Regulatory T lymphocytes (Treg) participate in the maintenance of immune system homeostasis by ensuring tolerance to self antigens. Within TME, Treg inhibit anti-tumor T cell activity and potentiate tumor proliferation. The latter, by specifically recognizing tumor antigens, block the activity of effector T lymphocytes directed against tumor cells. Thus, an increase in circulating Treg concentrations and in TME is a poor prognostic factor, especially in NSCLC.

Gemcitabine chemotherapy is commonly used in the management of NSCLC. Recent data show that gemcitabine decreases Treg activity and regulates levels of anti-inflammatory TME cytokines such as IL10, TGF-β and interferon-Ɣ.

The hypothesis of this study is that the decrease in Treg blood concentration by catch-up chemotherapy restores sensitivity to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients treated with immune checkpoint inhibitor alone or in combination with chemotherapy in 1st or 2nd line
* Patient with locally advanced or metastatic Non-Small-Cell Lung Cancer, or bladder cancer or Ear Nose Throat cancer
* Maximum delay of 2 months between ICI and chemotherapy

Exclusion Criteria:

* Symptomatic brain metastases
* Corticotherapy > 10 mg/day
* Active auto-immune disease
* Oncogenic addiction
* Data processing objection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients receiving chemotherapy alone after immunotherapy for NSCLC or bladder cancer or ENT cancer.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood concentration of regulatory T-lymphocytes (Treg) at 6 months | Baseline, 3 months and 6 months
  Blood concentrations will be measured at specific times
Change from baseline blood concentration of lymphocyte populations T, B, NK, CD4+ and CD8+ (effector T-lymphocytes (Teff) included) at 6 months | Baseline, 3 months and 6 months
  Blood concentrations will be measured at specific times

SECONDARY OUTCOMES:
Change from baseline blood concentration of anti-inflammatory cytokines at 6 months | Baseline, 3 months and 6 months
  Blood concentrations will be measured at specific times
Assess correlation between blood concentration of Treg, blood concentration of Teff and blood concentration of anti-inflammatory cytokines | Baseline, 3 months and 6 months
Determination of PDL1 status | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Medical oncology department, University Hospital, Tours, Tours
  - Pneumology department, University Hospital, Tours, Tours